CLINICAL TRIAL: NCT01670149
Title: A Randomised Placebo Controlled Trial of "Follow on" Rifaximin for the Prevention of Relapse of Clostridium Associated Diarrhoea
Brief Title: Rifaximin for Preventing Relapse of Clostridium Associated Diarrhoea
Acronym: RAPID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12072; 2012-003205-10 (EudraCT Number)
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; Diarrhoea; Rifaximin
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Identical looking tablet
  Interventions: Drug: Placebo
- Rifaximin , Xifaxanta™ (Active Comparator): 2 weeks of Rifaximin 400mg thrice daily then 2 weeks of Rifaximin 200mg thrice daily Modified Xifaxanta™ (rifaximin film-coated tablet) manufactured by Alfa Wasermann (AW),
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Tablets
  Other Names: Xifaxanta™
  Arms: Rifaximin , Xifaxanta™
Drug: Placebo — Tablets
  Arms: Placebo

SUMMARY:
Clostridium difficile associated diarrhoea is an important cause of morbidity in patients treated with antibiotics, especially in hospital. Clinical relapse occurs after up to 30% of initially successful treatments for colitis. Preliminary reports suggest that Rifaximin, a poorly absorbed antibiotic used to treat travellers diarrhoea can prevent relapse. We plan to carry out a randomised placebo controlled trial to test the hypothesis that Rifaximin given in a reducing dose over 4 weeks after successful treatment will reduce the relapse rate.

DETAILED DESCRIPTION:
Aims i) To examine efficacy of a follow-on course of Rifaximin given after a successful initial course of standard treatment, in the prevention of relapse in C. difficile associated diarrhoea (CDAD).

ii) To examine changes in faecal microbiota in patients given Rifaximin vs. Placebo.

Treatment 4 weeks treatment with Rifaximin or Placebo tablets. Tapering dose starting with 2 x 200mg tablets three times a day (total = 1.2g per day) for the 1st 2 weeks, reduced to 1 x 200mg tablet three times a day (total = 0.6g per day) for the 2nd 2 weeks.

Primary endpoint: The difference in % relapse between Rifaximin and placebo at 12 weeks

ELIGIBILITY:
Inclusion criteria:

1. Men / Women aged 18 and over (We will also include those adults who lack mental capacity for whom we have a legal representative)
2. Successful treatment of clinically diagnosed CDAD using standard therapy (metronidazole or vancomycin given according to standard local hospital guidelines).

Exclusion criteria:

1. Woman of child bearing potential and not willing to use at least one highly effective contraceptive method throughout the study
2. Male with spouse/partner of child bearing potential and not willing to use condoms
3. Pregnant or breast feeding
4. Unable to swallow tablets
5. Life expectancy of <4 weeks
6. Hypersensitivity to the active substance, to any rifamycin (e.g. rifampicin or rifabutin) or to any of its excipients (Tablet core: Sodium starch glycolate type A, glycerol distearate, colloidal anhydrous, silica, talc and microcrystalline cellulose. Tablet coating: hypromellose, titanium dioxide (E171), disodium edentate, propylene glycol and red iron oxide E172)
7. >5 days post standard therapy (metronidazole or vancomycin) for clinically diagnosed CDAD
8. Taking ciclosporin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2012-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Difference in % relapse between Rifaximin and placebo at 12 weeks | 12 weeks
  The difference in % relapse between Rifaximin and placebo at 12 weeks

SECONDARY OUTCOMES:
Proportion relapsed, re-hospitalisation and bowel symptoms | 12 weeks - 6 months
  Secondary endpoints:
  Clinical:
  1. Proportion with relapse of CDAD within 6 months
  2. Proportion re-hospitalised for CDAD within 6 months
  3. Length of in-hospital stay following start of treatment
  Exploratory:
  1. Stool frequency and consistency during 12 weeks after start of treatment
  2. Microbiological assessments

CONTACTS AND LOCATIONS:
Overall Officials: Aida Jawhari, MD, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham Clinical Trials Unit (NCTU), Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Major G, Bradshaw L, Boota N, Sprange K, Diggle M, Montgomery A, Jawhari A, Spiller RC; RAPID Collaboration Group. Follow-on RifAximin for the Prevention of recurrence following standard treatment of Infection with Clostridium Difficile (RAPID): a randomised placebo controlled trial. Gut. 2019 Jul;68(7):1224-1231. doi: 10.1136/gutjnl-2018-316794. Epub 2018 Sep 25. PMID 30254135
- [Derived] Stevenson EC, Major GA, Spiller RC, Kuehne SA, Minton NP. Coinfection and Emergence of Rifamycin Resistance during a Recurrent Clostridium difficile Infection. J Clin Microbiol. 2016 Nov;54(11):2689-2694. doi: 10.1128/JCM.01025-16. Epub 2016 Aug 24. PMID 27558181
- See also: Summary results EU Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2012-003205-10/results